CLINICAL TRIAL: NCT05182710
Title: Preparing for the Stress of Resuscitation: A Randomised Control Trial of Simulation-based Stress Inoculation Training for UK Medical Professionals
Brief Title: Simulation-based Stress Inoculation Training Study for UK Medical Professionals
Acronym: SITS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021.RCHT.86
Record Dates: First submitted 2021-11-08; First posted 2022-01-10 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Stress; Stress, Psychological; Stress, Job
Keywords: Stress Inoculation Training; SIT; NHS; Doctor; Resuscitation; Simulation; Medical Education
MeSH Terms: conditions — Stress, Psychological; Occupational Stress

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which of the two interventions (training modules) is being assessed.
  Those facilitating simulations will also be blinded. Those assessing over-all effectiveness of resuscitation will be blinded to which arm participants are in
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Inoculation Training (Experimental): Intervention Arm
  Interventions: Behavioral: Stress Inoculation Training
- Alternative Training (Active Comparator): Best practice/control
  Interventions: Behavioral: Alternative Training

INTERVENTIONS:
Behavioral: Stress Inoculation Training — The SIT programme/intervention will involve
  1. 30 minute educational phase of preparatory information to allow participants to conceptualise the types of stressors they are likely to face and the role of stress on performance
  2. 30 minutes of skills acquisition which will involve discussion of and teaching participants techniques to reduce stress in simulated resuscitation events
  3. Inoculation through the application of acquired skills in 1-2 resuscitation scenarios
  Arms: Stress Inoculation Training
Behavioral: Alternative Training — 1. 30 minutes of teaching on management of a drowning patient (in order that both control and intervention perceive they have had teaching of the same length as the other group)
  2. 1-2 resuscitation simulation events (same scenario and tasks as in the intervention group)
  Arms: Alternative Training

SUMMARY:
This study is to assess for the effectiveness of a Simulation-Based Stress Inoculation Training (SIT) Programme for junior doctors and physicians associates. It was well known that clinical practice can be stressful, particularly resuscitation events. When practitioners are stressed, they become less clinically effective. However, this is little in the way of training on how to manage acute stress in the workplace.

Stress Inoculation Training is established in military and sports training but is yet to be researched fully in junior doctors or physicians associates. By integrating a SIT programme into regular simulation training, the study aims to assess whether it helps with managing stress and performing better resuscitation. This assessment will be via questionnaire, heart rate monitors and judgement of clinical performance.

The study will be open to junior doctors and physicians associates who are currently practicing at the Royal Cornwall Hospital Trust and will take place in the Simulation Suite over a 6 month period.

Results will be prepared for publication and circulated among participants

DETAILED DESCRIPTION:
This study is a randomised control trial design. The study aim is to obtain 40 participants of varied roles, all healthcare professionals at the NHS RCHT. Participants will be asked to sign up to a session run in regular working hours at the RCHT simulation suite. If participants wish to take part in the study, after being consented to the project, they will be randomised to either the intervention arm or control arm.

Best practice/control is as follows

1. 30 minutes of teaching on management of a drowning patient (or similar topic, in order that both control and intervention perceive they have had teaching of the same length as the other group)
2. 1-2 resuscitation simulation events (same scenario and tasks as in the intervention group)

The SIT programme/intervention will involve

1. 30 minute educational phase of preparatory information to allow participants to conceptualise the types of stressors they are likely to face and the role of stress on performance
2. 30 minutes of skills acquisition which will involve teaching participants techniques to reduce stress in simulated resuscitation events
3. Inoculation through the application of acquired skills in 1-2 resuscitation scenarios

All participants will be asked to complete a State-Trait Anxiety Inventory (STAI) questionnaire both prior to and immediately after the end of each scenario All participants will have their heart rates monitored throughout the session with timings correlated against stressors and application of stress reduction techniques

All participants will have the same set of scenarios involving the same tasks. Performance at individual tasks (such as cannulation, guide wire fitting, ECG interpretation, ABG interpretation, recalling allergies, noticing equipment failure) and overall performance will be assessed by an independent, blinded assessors according to a pre-determined score scheme using video footage of each scenario

Scenarios will be facilitated by blinded researchers. These facilitators will be members of the simulation team. For the duration of the session, they will be based on the simulation room and not take part in the training modules. They will not be aware if simulation participants are part of the control or intervention group. They will be tasked with running the simulation scenario with consistency across participants.

Data analysis will include using MSExcel to test for statistically significant differences in biomarkers, self-reported scores and independent, blinded assessor scores. All results will be identified by using an anonymous code for each participant which will reference only their job role and whether they are in the intervention or control group* (badges will be worn by participants for identification).

*this may have to be done via a code so independent assessors watching the videos do not know

Data, including videos of the simulation session, photocopies of the STAI questionnaire and transcribed heart rate values will be stored anonymously on the RCHT server and not copied across to any personal or other devices. It will only be accessed my primary researchers. Videos will be stored in a separate folder which the independent assessor will have access to and photocopies of their mark schemes will be uploaded to the RCHT server also. All paper forms will be shredded using the hospital's existing system for disposal of confidential waste

ELIGIBILITY:
Inclusion Criteria:

* Any medical professional (junior doctors or physicians associates) currently working part/full time at RCHT
* A current licence to practice
* Willing to consent to participate in the study

Exclusion Criteria:

* Anyone taking a medication which modifies heart rate (eg betablockers)
* Unwilling to consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | 10 minutes during simulation scenario
  Difference in heart rate variability during simulated resuscitation events (objective measure)
State-Trait Anxiety Inventory Difference | STAI takes about 1 minute to complete and participants will be asked to complete it 5 minutes before and 5 minutes after simulation event
  Difference in State-Trait Anxiety Inventory (STAI) scores before and after resuscitation events (subjective measure)

SECONDARY OUTCOMES:
Motor Task Capacity | Participants will be given 1 minute to complete this task during the simulation event, before being asked to move on and continue the scenario
  Difference in time (seconds) taken to perform a fine motor task. This task will involve insertion of catheter onto guide wire during simulated resuscitation event
Cognitive Capacity | Participants will be given 1 minute to complete this task during the simulation event, before being asked to move on and continue the scenario
  Difference in time (seconds) taken to perform a cognitive task. This task will involve interpreting an Electrocardiogram (ECG) or Arterial Blood Gas (ABG) during simulated resuscitation event
Situational Awareness Capacity | Participants will be given 1 minute to complete this task during the simulation event, before being asked to move on and continue the scenario
  Difference in time (seconds) taken to demonstrate situational awareness. This task will involve participants recognising a device failure such as detachment of ECG leads and loss of ECG trace during simulated resuscitation event
Effectiveness of Resuscitation | An independent assessor will review the videos of simulation events within 2 months of the simulation event. Each simulation should last around 10 minutes
  Difference in overall performance as assessed by independent expert. The expert will be asked to rank the overall effectiveness of the resuscitation on a scale of 1 to 10 where 1 is entirely ineffective resuscitation and 10 is entirely effective resuscitation

OTHER OUTCOMES:
Self-reported stress in real resuscitation events | 5 minute questionnaire conducted between 1 and 3 months following training and simulation event
  Difference in self reported stress at work after simulated resuscitation event. Participants will be asked to rank their level of stress/anxiety on a scale of 1 to 10 in three scenarios: anticipation of a real resuscitation event, during a real resuscitation event, after a real resuscitation event

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Connolly, MBChB, FRSA, Study Chair — National Health Service (NHS)
Locations (1):
- Post-Graduate Centre, Royal Cornwall Hospital NHS Trust, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared generally. Individual level data will only be shared within the primary research team and only when strictly necessary